CLINICAL TRIAL: NCT05688670
Title: Pain Control With Regional Anesthesia Following Pediatric Cardiac Surgery: A Randomized Double-Blinded Pilot Study
Brief Title: Regional Anesthesia Following Pediatric Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Society of Pediatric Anesthesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00111671
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Atrial Septal Defect; Ventricular Septal Defect; Pain, Procedural
Keywords: Regional anesthesia
MeSH Terms: conditions — Heart Septal Defects, Atrial; Heart Septal Defects, Ventricular; Pain, Procedural | interventions — Anesthesia, Conduction; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regional Anesthesia (Active Comparator): Ultrasound guided blocks
  Interventions: Procedure: Regional Anesthesia; Drug: Ropivacaine 0.2% Injectable Solution
- Wound Infiltration (Active Comparator): Surgeon-delivered wound infiltration
  Interventions: Procedure: Wound infiltration; Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Procedure: Regional Anesthesia — Bilateral pecto-intercostal fascial plane block (PIFB) and unilateral rectus sheath block (RSB) with Ropivacaine 0.2%
  Arms: Regional Anesthesia
Procedure: Wound infiltration — Surgeon-delivered wound infiltration with Ropivacaine 0.2%
  Arms: Wound Infiltration
Drug: Ropivacaine 0.2% Injectable Solution — Ropivacaine 1.5 mL/kg will be used for both interventions

SUMMARY:
The purpose of this study is to evaluate pain control following pediatric cardiac surgery with the use of local anesthesia via an ultrasound guided regional anesthetic technique compared with surgeon delivered wound infiltration.

DETAILED DESCRIPTION:
This is a single center, randomized, double blind investigation which will compare postoperative pain control indices, functional recovery metrics and patient/parental satisfaction for pediatric patients receiving an ultrasound guided regional anesthetic versus surgeon delivered wound infiltration in children undergoing primary atrial and ventricular septal defect repairs. Surgical and anesthesia care, with the exception of the technique of local anesthetic administration, are not altered for study purposes. Subjects are randomized 1:1 to either bilateral Pecto-Intercostal Fascial Block and unilateral Rectus Sheath Block or infiltration of the wound through the perioperative period. Both interventions will use an equal volume of Ropivacaine 0.2% based on weight. Exploratory data will be collected for up to 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Children less than 18 years old
2. Presenting for primary atrial septal defect or ventricular septal defect repair
3. Informed consent / assent provided

Exclusion Criteria:

1. Patients on opioid therapy at the time of surgery
2. History of sternotomy
3. Planned postoperative intubation
4. Current diagnosis of a chronic pain syndrome.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2025-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Einhorn, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Regional Anesthesia: Ultrasound guided blocks Regional Anesthesia: Bilateral pecto-intercostal fascial plane block (PIFB) and unilateral rectus sheath block (RSB) with Ropivacaine 0.2% Ropivacaine 0.2% Injectable Solution: Ropivacaine 1.5 mL/kg will be used for both interventions
- Wound Infiltration: Surgeon-delivered wound infiltration Wound infiltration: Surgeon-delivered wound infiltration with Ropivacaine 0.2% Ropivacaine 0.2% Injectable Solution: Ropivacaine 1.5 mL/kg will be used for both interventions
Period: Overall Study
Arm/Group | Regional Anesthesia | Wound Infiltration
Started | 26 | 26
Completed | 24 | 18
Not Completed | 2 | 8
Not completed — Change in surgery plan | 1 | 4
Not completed — Inability to extubate | 1 | 2
Not completed — Day of surgery cancellation | 0 | 1
Not completed — Reintubated on PCICU arrival | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed data collection for the primary and secondary outcomes (up to 48 hours after surgery) are reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regional Anesthesia | Wound Infiltration | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3 [0.3 to 10] | 3 [0.3 to 9] | 3 [0.3 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 19 | 15 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 18 | 11 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Opioid Medications Administered
Description: Postoperative opioid medication expressed in morphine equivalents per kilogram
Time Frame: Up to 12 hours after surgery
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: MME/kg
Arm/Group | Regional Anesthesia | Wound Infiltration
Number analyzed (Participants) | 24 | 18
MME/kg | 0.44 (0.19) | 0.83 (0.39)
Statistical Analysis 1: Comparison: Regional Anesthesia vs Wound Infiltration; Test type: Superiority; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.59 to -0.18]

2. Secondary Outcome: Total Amount of Opioid Medications Administered
Description: Postoperative opioid medication expressed in morphine equivalents per kilogram
Time Frame: 12-24 hours after surgery; 24-48 hours after surgery; 12-48 hours hours after surgery
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: MME/kg
Arm/Group | Regional Anesthesia | Wound Infiltration
Number analyzed (Participants) | 24 | 18
MME/kg
  12-24 hours after surgery | 0.29 (0.19) | 0.35 (0.24)
  24-48 hours after surgery | 0.23 (0.22) | 0.39 (0.39)
  12-48 hours hours after surgery | 0.52 (0.32) | 0.74 (0.56)
Statistical Analysis 1: Comparison: Regional Anesthesia vs Wound Infiltration; 12-24 hour postoperative opioid use; Test type: Superiority; p = 0.41, t-test, 2 sided; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.20 to 0.08]
Statistical Analysis 2: Comparison: Regional Anesthesia vs Wound Infiltration; 24-48 hour postoperative opioid use; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.37 to 0.06]
Statistical Analysis 3: Comparison: Regional Anesthesia vs Wound Infiltration; 12-48 hours hours after surgery; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.52 to 0.09]

3. Secondary Outcome: Total Amount of Opioid Medications Administered
Description: Postoperative opioid medication expressed in morphine equivalents per kilogram
Time Frame: Up to 48 hours after surgery
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: MME/kg
Arm/Group | Regional Anesthesia | Wound Infiltration
Number analyzed (Participants) | 24 | 18
MME/kg | 0.95 (0.40) | 1.57 (0.75)
Statistical Analysis 1: Comparison: Regional Anesthesia vs Wound Infiltration; Test type: Superiority; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.02 to -0.22]

4. Secondary Outcome: Postoperative Pain Intensity AUC
Description: Cumulative burden of pain over time was assessed using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale. Scores range from 0-10, with higher scores indicating greater pain.
Time Frame: 48 hours
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: FLACC pain score (0-10)*hours
Arm/Group | Regional Anesthesia | Wound Infiltration
Number analyzed (Participants) | 24 | 18
FLACC pain score (0-10)*hours | 45.0 (26.8) | 94.5 (55.7)
Statistical Analysis 1: Comparison: Regional Anesthesia vs Wound Infiltration; Test type: Superiority; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = -49.5, 95% CI 2-sided [-78.9 to -20.1]

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Regional Anesthesia | Wound Infiltration
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT05688670/Prot_SAP_000.pdf